CLINICAL TRIAL: NCT02251392
Title: Evaluation of Therapeutic Efficacy in Use of Chamomila Gel, Chamomila Infuse and Urea in Patients With Breast or Head and Neck Cancer That Developed Radiodermatitis
Brief Title: Evaluation of Therapeutic Efficacy in Use of Chamomilla Gel, Chamomilla Infuse and Urea in Radiodermatitis
Acronym: ChamomillaTH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Brasilia (Other)
Collaborators: University of Washington (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, PAULA ELAINE DINIZ DOS REIS, PROFESSOR, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBrasilia
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Radiodermatitis
Keywords: chamomilla; matricaria; chamomile; chamomila; recutita; Breast Neoplasms; head and neck neoplasms; radiotherapy
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chamomila recutita Gel (Experimental): Experimental Group 1 - patients will apply the gel since the begging of radiodermatitis, three times a day. The dose is being determined in a Phase II study that is being conducted. Topical application of gel is going to occur concomitantly to the initiation of radiodermatitis and will be follow up until the cure of it.
  Interventions: Other: Chamomila recutita Gel
- Chamomila recutita Infuse 2,5% (Experimental): Experimental Group 2 - patients will apply the infuse since the begging of radiodermatitis, three times a day. The dose of 2,5% was determined before in a Phase II study. Radiodermatitis grade and intensity is going to be evaluated. Topical application of the infuse is going to occur concomitantly to the initiation of radiodermatitis and will be follow up until the cure of it.
  Interventions: Other: Chamomila recutita Infuse
- Urea cream based (Active Comparator): Control Group - usual care to treat radiodermatitis, patients will apply the infuse since the begging of radiodermatitis, three times a day. Radiodermatitis grade and intensity is going to be evaluated. Topical application of urea is going to occur concomitantly to the initiation of radiodermatitis and will be follow up until the cure of it.
  Interventions: Drug: Urea cream based

INTERVENTIONS:
Other: Chamomila recutita Gel — Gel formulated with active principles from Chamomilla recutita which dose is being determined in a dose-response curve
  Other Names: Chamomile Gel, Chamomila recutita gel
  Arms: Chamomila recutita Gel
Other: Chamomila recutita Infuse — chamomila infuse in a concentration of 2,5% already determined in a dose response curve
  Other Names: Chamomile Infuse, Chamomila recutita infuse
  Arms: Chamomila recutita Infuse 2,5%
Drug: Urea cream based — Urea is already using to treat radiodermatitis when it starts to occur, so it will be the usual care
  Other Names: Urea cream
  Arms: Urea cream based

SUMMARY:
This study aims to evaluate therapeutics interventions in radiodermatitis in patients with breast or head and neck cancer. The data collect is going to begin after determining the better dose in a dose-response curve that is being conduct now in the same institution. To evaluate the skin reaction will be applied scale of the Radiation Therapy Oncology Group (RTOG) - Acute Radiation Morbidity Scoring Criteria, Common Terminology Criteria for Adverse Events (CTCAE) and Radiation-Induced Skin Reaction Assessment Scale (RISRAS).

DETAILED DESCRIPTION:
Hypothesis:

Chamomila gel is more effective than urea (usual care); Chamomila infuse is more effective than urea (usual care); Chamomila gel is more effective than chamomila infuse; Chamomila infuse is more effective than chamomila gel; Chamomila gel is as effective than urea (usual care); Chamomila infuse is as effective than urea (usual care); Chamomila gel is as effective than chamomila infuse; Chamomila infuse is as effective than chamomila gel.

ELIGIBILITY:
Inclusion Criteria:

Being an adult, over the age of 18 years old; Owning diagnosis of breast or head and neck cancer; Being first referred to the radiotherapy protocol; Presenting radiodermatitis grades 1 or 2, second RTOG score, in the place where is receiving radiation therapy; No history of previous hypersensitivity reaction to chamomile or any plant of the Asteraceae or Compositae family or Urea; Demonstrate understanding to continue the intervention in their home environment when necessary.

Exclusion Criteria:

Medical prescription, during the process of data collection, some kind of intervention to prevent radiodermatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the severity of radiodermatitis, according to the RTOG score. | 5 weeks
  This outcome is going to be evaluated weekly by the analisys of the signs and symptoms of radiodermititis ant the RTOG score

SECONDARY OUTCOMES:
Radiation Dose | 5 weeks
  radiation total dose and fraction
Radiodermititis Cure | 8 weeks
  The time that pacient don´t have more the radiodermititis
Time to reduce the severity of radiodermatitis | 5 weeks
  This outcome is going to be evaluated weekly by the analisys of the time of reduce the signs and symptoms of radiodermititis ant the RTOG score

CONTACTS AND LOCATIONS:
Overall Officials: Elaine B Ferreira, Nurse, Principal Investigator — University of Brasilia; Priscila MS Bontempo, Nurse, Principal Investigator — University Hospital of Brasilia; Marcia A Ciol, Biostatistcs, Study Director — University of Washington; Karine RM Silva, Nurse, Study Chair — University of Brasilia; Carlos J Sacramento, Nurse, Study Chair — University of Brasilia; Paula ED Reis, PhD, Nurse, Study Director — University of Brasilia; Samuel R Avelino, MP, Principal Investigator — University Hospital of Brasilia; Leandro X Cardoso, Physics, Study Chair — University of Brasilia; Luis FO Silva, MP, Study Chair — University Hospital of Brasilia

REFERENCES:
- [Background] Reis PE, Carvalho EC, Bueno PC, Bastos JK. Clinical application of Chamomilla recutita in phlebitis: dose response curve study. Rev Lat Am Enfermagem. 2011 Jan-Feb;19(1):3-10. doi: 10.1590/s0104-11692011000100002. PMID 21412623